CLINICAL TRIAL: NCT06863558
Title: Reduction of Edema With a Specialized Cocktail for Ultra-early Management in Intracerebral Hemorrhage
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCUE-ICH
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPA Intervention Group (Experimental): Participants in this group will receive a pharmacological cocktail (PPA) for five days in addition to standard medical treatment for acute ischemic stroke. The regimen includes terazosin or urapidil, and propranolol or esmolol, with individualized blood pressure management. The specific protocol is as follows:
  * Terazosin (no less than 1 mg orally or via nasogastric tube, nightly) or Urapidil (100 mg in 30 mL saline, IV infusion at no less than 2 mL/h)
  * Propranolol (10 mg orally or via nasogastric tube, three times daily) or Esmolol (1 g in 40 mL saline, IV infusion at no less than 2 mL/h; use for no more than 48 hours. Beyond 48 hours, switch to Propranolol)
  Interventions: Drug: PPA Intervention
- Standard Treatment Group (No Intervention): Participants in this group will receive standard medical treatment for acute ischemic stroke without the PPA intervention. This includes appropriate supportive care, blood pressure management according to clinical guidelines, and symptomatic treatment as required.

INTERVENTIONS:
Drug: PPA Intervention — Participants in this group will receive a pharmacological cocktail (PPA) for five days in addition to standard medical treatment for acute ischemic stroke. The regimen includes terazosin or urapidil, and propranolol or esmolol, with individualized blood pressure management. The specific protocol is as follows:
  * Terazosin (no less than 1 mg orally or via nasogastric tube, nightly) or Urapidil (100 mg in 30 mL saline, IV infusion at no less than 2 mL/h)
  * Propranolol (10 mg orally or via nasogastric tube, three times daily) or Esmolol (1 g in 40 mL saline, IV infusion at no less than 2 mL/h; use for no more than 48 hours. Beyond 48 hours, switch to Propranolol)
  Arms: PPA Intervention Group

SUMMARY:
Intracerebral hemorrhage (ICH) is a severe stroke subtype with high mortality and disability rates, often worsened by perihematomal edema (PHE), which increases intracranial pressure and leads to poor outcomes. Preclinical studies suggest that a pharmacological cocktail (PPA) may help reduce cerebral edema by modulating potassium balance, preserving aquaporin-4 expression, and enhancing lymphatic drainage.

This multicenter, randomized controlled trial (RCT) aims to evaluate the safety and efficacy of PPA in ICH patients. A total of 58 patients with supratentorial ICH (≥3 mL hematoma volume) who are not undergoing surgical evacuation will be randomized to receive either PPA therapy or standard treatment. The primary outcome is the change in cerebral edema volume at 5-7 days, assessed by CT imaging. Secondary outcomes include 90-day functional outcomes (mRS), need for decompressive craniectomy, and safety assessments. This study seeks to explore PPA as a potential treatment strategy for cerebral edema in ICH patients.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is a severe subtype of stroke, accounting for 15-20% of all strokes. Compared to ischemic stroke, ICH has a higher mortality and disability rate, with its incidence steadily rising worldwide, imposing a substantial burden on families and healthcare systems. A key factor contributing to poor prognosis in ICH is perihematomal edema (PHE), which rapidly progresses during the acute phase, leading to increased intracranial pressure (ICP), brain tissue displacement, and potential brain herniation. Even in patients who survive the acute phase, persistent cerebral edema can cause long-term neurological deficits and impair quality of life. Therefore, effective management of cerebral edema is critical for improving outcomes in ICH patients.

Preclinical studies suggest that a pharmacological cocktail (PPA), consisting of adrenergic antagonists, may help reduce cerebral edema by modulating extracellular potassium homeostasis, maintaining aquaporin-4 (AQP-4) expression, and enhancing lymphatic drainage. In both traumatic brain injury and ischemic stroke models, PPA has shown potential in alleviating cerebral edema and improving neurological recovery. Based on these findings, this multicenter, randomized controlled trial (RCT) aims to evaluate the safety and efficacy of PPA in reducing cerebral edema in ICH patients.

The study will enroll 58 patients diagnosed with supratentorial ICH (≥3 mL hematoma volume) who are not undergoing surgical evacuation. Participants will be randomly assigned to receive PPA therapy or standard treatment. The primary outcome is change in cerebral edema volume at 5-7 days, assessed by CT imaging. Secondary outcomes include functional outcomes at 90 days (mRS), need for decompressive craniectomy, incidence of hypotension, and adverse events. This study aims to explore PPA as a novel pharmacological approach for managing cerebral edema in ICH, potentially improving patient prognosis and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of supratentorial intracerebral hemorrhage (ICH)
* Symptom onset within 3 days (≤72 hours) before randomization
* Baseline CT-confirmed hematoma volume ≥3 mL
* Not scheduled for hematoma evacuation surgery (either not indicated or declined by the patient/family)
* Written informed consent obtained from the patient or legally authorized representative

Exclusion Criteria:

* Baseline brain herniation or severe hypotension (SBP <90 mmHg)
* Contraindications to PPA medications (terazosin, urapidil, esmolol, propranolol), such as asthma or severe bradycardia
* Severe comorbidities that may interfere with efficacy assessment or pose a high safety risk (e.g., end-stage organ failure, advanced malignancy)
* Presence of secondary causes of ICH (e.g., arteriovenous malformation, aneurysm rupture, hemorrhagic transformation of ischemic stroke)
* Pregnancy or lactation
* Participation in another interventional trial that may influence study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral Edema Volume at 5-7 Days | Baseline and 5-7 days post-treatment
  The primary outcome of this study is the change in cerebral edema volume, as assessed by non-contrast CT imaging at baseline (pre-treatment) and 5-7 days after treatment initiation. Edema volume will be quantified using standardized imaging analysis techniques. The difference in cerebral edema volume between the PPA intervention group and the standard treatment group will be compared to evaluate the efficacy of the pharmacological cocktail in reducing brain swelling.

SECONDARY OUTCOMES:
90-Day Functional Outcome (Modified Rankin Scale, mRS) | 90 days post-treatment
  Functional outcomes will be assessed using the modified Rankin Scale (mRS) at 90 days post-treatment, mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Incidence of Hypotension During the Treatment Period | Time Frame: During the 5-day treatment period
  The occurrence of clinically significant hypotension (defined as systolic blood pressure <90 mmHg) will be monitored throughout the intervention period. The frequency, severity, and need for medical intervention will be compared between the two study groups.
Change in Hematoma Volume | 5-7 days post-treatment
  Assessment of hematoma volume on CT imaging at baseline and 5-7 days post-treatment to evaluate any changes in bleeding size.
Need for Decompressive Craniectomy | Up to 7 days
  The proportion of patients who require decompressive craniectomy due to increased intracranial pressure or neurological deterioration.
Mortality at 90 Days | 90 days post-treatment
  All-cause mortality will be recorded and compared between the PPA intervention and standard treatment groups to evaluate the impact of the intervention on survival.
Incidence of Serious Adverse Events (SAEs) | Up to 90 days post-treatment
  All serious adverse events (SAEs), including cardiovascular complications, major bleeding, and severe drug reactions, will be recorded and compared between groups.

IPD SHARING:
Plan to Share IPD: Undecided